CLINICAL TRIAL: NCT00817895
Title: Clinical Randomized Control Trial of Intraoperative Implanting Chemotherapeutic Drugs Sustained Release Following Resection of Hepatocellular Carcinoma Against Postoperative Short-term Recurrence
Brief Title: Intraoperative Chemotherapy Against Hepatocellular Carcinoma Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EHBH-RCT-2008-010
Record Dates: First submitted 2009-01-04; First posted 2009-01-07 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; liver resection; intraoperative chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5-FU+Cisplatin (Experimental): 50 HCC patients will be implanted 600mg sustained released 5-FU and 60mg sustained released cisplatin into liver incisal margin after tumor is resected.
  Interventions: Drug: sustained released 5-FU and sustained released cisplatin; Procedure: TACE
- 5-FU (Active Comparator): 50 HCC patients will be implanted 600mg sustained released 5-FU into liver incisal margin after tumor is resected.
  Interventions: Drug: sustained released 5-FU; Procedure: TACE
- control (Experimental)
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: sustained released 5-FU and sustained released cisplatin — 600mg sustained released 5-FU and 60mg sustained released cisplatin will be implanted into liver incisal margin after tumor is resected.
  Other Names: 5-FU+Cisplatin group
  Arms: 5-FU+Cisplatin
Drug: sustained released 5-FU — 600mg sustained released 5-FU will be implanted into liver incisal margin after tumor is resected.
  Other Names: 5-FU group
  Arms: 5-FU
Procedure: TACE — All patients will accept TACE one month after tumor was resected.
  Other Names: Postoperative TACE

SUMMARY:
Hepatectomy is still the most important treatment for HCC.High recurrence rate mostly influence it's prognosis, especially for the patient with tumor >5cm, multiple tumor and who cannot accept R0 resection.Our retrospective study showed sustained released 5-FU implanted into the liver incisal margin after tumor was resected could reduce the recurrence rate of HCC after liver resection.According to this, we proceed this RCT to prospectively observe the effect of sustained released 5-FU,and we also want to know whether combined with sustained released cisplatin will get better effect in preventing the tumor recurrence,especially in short time after liver resection.

DETAILED DESCRIPTION:
150 HCC patients with tumor >5cm, multiple tumor and who cannot accept R0 resection will be randomized divided into 3 groups. Group A (50 cases) will be implanted 600mg sustained released 5-FU into liver incisal margin after tumor is resected. Group B (50 cases) will be implanted 600mg sustained released 5-FU and 60mg sustained released cisplatin. Group C (50 cases) will be the controlled one which will not be implanted any chemotherapeutic drugs. All patients will accepted TACE 30 days after liver resection. We will follow up all patients until they are dead or missed connected. Related adverse reaction will be recorded. Total survival time (TST) and disease free survival time (DFST) will be calculated too. At the end of the study we will compare the difference of adverse reaction, complication, TST and DFST between the 3 groups. According to the result we will estimate these drugs' antitumor effect and safety.

ELIGIBILITY:
Inclusion Criteria:

1. tumor >5cm;
2. multiple tumor located in one liver lobe;
3. margin of tumor is not clear;
4. cutting edge to tumor <1cm;
5. portal vein branch invasion;
6. without extra-liver metastasis;
7. patient's liver function and condition is able to accept hepatectomy.

Exclusion Criteria:

1. single tumor <=5cm;
2. multiple tumor located more than in one liver lobe;
3. margin of tumor is clear;
4. cutting edge to tumor >=1cm;
5. portal vein stem invasion
6. extra-liver metastasis;
7. patient's liver function and condition cannot accept hepatectomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
disease free survival | 2 years

SECONDARY OUTCOMES:
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD., Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China